CLINICAL TRIAL: NCT06253949
Title: Evaluation of Clinical and Oncological Outcomes After High and Low Ligation of Inferior Mesenteric Artery in Elective Left-sided Colon and Rectal Cancer
Brief Title: Compare Outcomes After High and Low Ligation of Inferior Mesenteric Artery in Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ramadan Mohamed, Assistant Lecturer of General Surgery Faculty of Medicine, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-01-01MD
Record Dates: First submitted 2024-02-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer
Keywords: colon cancer; high tie; low tie; inferior mesenteric artery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high tie ligation of inferior mesenteric artery (Active Comparator): Group A patients of elective operable colorectal cancer : high tie group
  Interventions: Procedure: ligation of inferior mesenteric artery in colorectal cancer
- low tie ligation of inferior mesenteric artery (Active Comparator): Group B patients of elective operable colorectal cancer : low tie group
  Interventions: Procedure: ligation of inferior mesenteric artery in colorectal cancer

INTERVENTIONS:
Procedure: ligation of inferior mesenteric artery in colorectal cancer — This study will include two groups of patients: group (A) and (B). In group (A), the inferior mesenteric artery will be ligated at its origin (high-tie), While in group (B), it will be ligated after the origin of the left colic artery (low-tie).

SUMMARY:
We aim comparing different outcomes between high and low tie ligation of inferior mesenteric artery in left colorectal cancer operable and elective surgeries.

DETAILED DESCRIPTION:
Colon cancer represents a significant clinical surgical burden, accounting for approximately 10% of all cancer cases. It is assumed that it is the second leading cause of cancer-related deaths worldwide. Surgery and chemotherapy are considered the main lines of treatment.

Left colonic and rectal cancers represent approximately two-thirds of all colorectal malignancies. The mainstay of treatment is surgical resection, including tumor removal with adequate safety margins with adequate lymphadenectomy.

Several lifestyle factors contribute to the development of colorectal cancer, such as a high intake of processed meats and low intake of fruits and vegetables, a sedentary lifestyle, obesity, smoking, and excessive alcohol consumption.

In colon and rectal cancer surgery, the approach toward the inferior mesenteric artery (IMA) has always been debated among surgeons regarding the "high tie" and "low tie" techniques.

According to the consensus statement of definitions of anorectal Physiology and Rectal Cancer of the American Society of Colon and Rectal Surgeons (ASCRS), a low tie of the IMA is meant as a ligation after the origin of the left colic artery. In contrast, the high tie a ligation of the IMA at its aortic root.

High ligation of the IMA for rectal and left colonic cancers may improve lymph node yield rate, thus facilitating more accurate tumor staging and better oncological outcomes. Several studies have shown the importance of lymph node dissection up to the root of the IMA in terms of better survival and precise staging. The high ligation also enables tension-free colonic anastomosis during low anterior resection. However, high ligation of the IMA has been known to decrease blood flow to the anastomosis, increasing the risk of anastomotic leak.

In contrast, the low-ligation technique allows for adequate blood supply to the colon proximal to the anastomotic stoma during low anterior resection that might prevent vascular inefficiency of the anastomotic marginal colic arteries and decrease the risk of anastomotic leak, especially in elderly patients.

On the other hand, low ligation limits the opportunity for lymph node clearance at the origin of the IMA. This incomplete lymphatic clearance may decrease survival while increasing the possibility of metastasis and cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Every elective patient diagnosed with left-side colon or rectal cancer will be included in our study.

Exclusion Criteria:

* Unfit patients with uncontrolled medical disease will be excluded. Patients with acute intestinal obstruction (emergency cases) and patients with extremes of age above 75 or pediatric ages will be excluded.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
anastomotic leakage | 2 weeks postoperative
  yes or no
hemorrhage | 2 weeks postoperative
  yes or no
rectal cancer-low anterior resection syndrome (LARS) | 2 weeks postoperative
  yes or no

SECONDARY OUTCOMES:
1-year overall survival | one year
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Mohamed, MD, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
not yet decided